CLINICAL TRIAL: NCT05806632
Title: Prognostic Relevance of Coagulation Activation in RIsk Assessment and Stratification in Reference to Patient Important Outcomes for Locally Advanced Breast Cancer: The ARIAS Trial
Brief Title: Prognostic Relevance of Coagulation Activation in RIsk Assessment and Stratification
Acronym: ARIAS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: RS1307/20
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Local Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Prognostic model — Risk assessment and risk stratification

SUMMARY:
Carcinogenesis and coagulation activation are closely related processes. In a previous study of coagulation activation in stage I-IIA breast cancer patients, we developed a prognostic model that includes coagulation activation biomarkers and demonstrated efficacy to in distinguish between risk categories and survival. Here, we propose a study useful for the validation of this prognostic model in an independent cohort of 108 patients with locally advanced breast cancer and indicated for neoadjuvant chemotherapy, followed by breast surgery. Within this study population, we will validate our prognostic model for risk assessment and risk stratification with respect to the following endpoints:

1. Complete pathological response rate to definitive breast surgery;
2. Rate of thromboembolic events.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal organ functions
* Cytologically/histologically proven breast cancer, stage IIB-IIIC
* Participants must not have prophylactic or therapeutic indications for anticoagulants.

Exclusion Criteria:

* Pregnacy
* Metastatic breast cancer
* Previous chemotherapy, hormone therapy, radiotherapy
* Previous malignancies or contralateral breast cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage IIB-IIIC breast cancer undergoing neoadjuvant chemotherapy (NACT), followed by breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | 30 months
  The study will mainly aim to validate the accuracy of previous developed prognostic model in distinguish between risk categories and probabilities of pathological complete response (pCR) detected in patients undergoing neoadjuvant chemotherapy (NACT) and breast surgery.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico Umberto I, Roma
  - Policlinico Agostino Gemelli, Roma
  - "Regina Elena" National Cancer Institute, Rome

IPD SHARING:
Plan to Share IPD: Undecided